CLINICAL TRIAL: NCT03458754
Title: Assessment of Exercise Capacity, Physical Activity, Pulmonary Function, Peripheric and Respiratory Muscle Strength, Respiratory Muscle Endurance in Patient With Peripheral Artery Disease
Brief Title: Maximal Exercise Capacity, Physical Activity and Respiratory Muscle Strength in Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof, Gazi University
Other Study IDs: Gazi University 9
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Exercise capacity; Physical activity; Respiratory muscle strength; Peripheric muscle strength
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Maximal exercise capacity will be assessed using cardiopulmonary exercise testing (CPET), functional exercise capacity using six minute stepper test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, depression using Beck depression inventory (Turkish version), life quality using SF-36 Health Survey (Turkish version), intermittent claudication using Walking Impairment Questionnaire (Turkish version)
- Healthy controls: Maximal exercise capacity will be assessed using cardiopulmonary exercise testing (CPET), functional exercise capacity using six minute stepper test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, depression using Beck depression inventory (Turkish version), life quality using SF-36 Health Survey (Turkish version), intermittent claudication using Walking Impairment Questionnaire (Turkish version)

SUMMARY:
The primary aim of the study is to evaluate the maximal and submaximal exercise capacity in patients with peripheral artery disease (PAD). The secondary aim of the study is assessment of physical activity level, respiratory function, peripheral and respiratory muscle strength, respiratory muscle endurance, depression, quality of life, intermittent claudication and cardiovascular risk factors in patients with PAD.

DETAILED DESCRIPTION:
Peripheral artery disease is characterized by reduced exercise capacity, physical activity level and intermittent claudication. The number of studies investigating maximal and submaximal exercise capacity and physical activity level in PAD is limited. There is also no study investigated pulmonary functions, respiratory muscle strength and endurance in this patient population. According to the sample size analysis 15 patients and 15 healthy individuals with similar demographic characteristics will be included the study. Patients and healthy individuals will be selected according to predetermined inclusion and exclusion criteria. The assessments will be completed in two days.Maximal exercise capacity will be assessed using cardiopulmonary exercise testing (CPET), functional exercise capacity using six minute stepper test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, depression using Beck depression inventory (Turkish version), life quality using SF-36 Health Survey (Turkish version), intermittent claudication using Walking Impairment Questionnaire (Turkish version)

ELIGIBILITY:
Inclusion Criteria:

Patients;

* Diagnosed with peripheral artery disease
* Ankle brachial index (ABI)≤ 1,5 or calcified vessel response
* Clinically stable and under standard medication patients will be included

Exclusion Criteria:

Patients with;

* Ischemic amputation
* Any pulmonary disease
* Unstable coronary artery disease
* Orthopedic and neurological problems
* Acute infection
* Myocardial infarction or major surgery in the last 3 months will be excluded

Healthy controls: Ages 18-80 years will be included

* With any diagnosed disease and smoking more than 10 packsyears will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 15 patients with PAD will be included in patients group and 15 healthy individuals will be included in control group
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | First day
  Cardiopulmonary exercise testing (Oxygen consumption measurement during test)

SECONDARY OUTCOMES:
Functional exercise capacity | Second day
  Six minute stepper test
Physical activity | Second day
  Multi sensor activity monitor
Pulmonary function | First day
  Spirometry
Respiratory muscle strength | First day
  Mouth pressure device
Peripheral muscle strength | Second day
  Hand held dynamometer
Respiratory muscle endurance | Second day
  Incremental threshold loading test
Depression | Second day
  Beck depression inventory (Turkish version)
Life quality | Second day
  SF-36 Health Survey (Turkish version)
Intermittent claudication | Second day
  Walking Impairment Questionnaire (Turkish version)

CONTACTS AND LOCATIONS:
Overall Officials: İnci Hazal Ayas, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Assoc. Prof, Study Director — Gazi University; Burcu Camcıoğlu, PhD, Principal Investigator — Gazi University; Dilek Erer, MD, Principal Investigator — Gazi University; Abdullah Özer, MD, Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Yenimahalle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leeper NJ, Myers J, Zhou M, Nead KT, Syed A, Kojima Y, Caceres RD, Cooke JP. Exercise capacity is the strongest predictor of mortality in patients with peripheral arterial disease. J Vasc Surg. 2013 Mar;57(3):728-33. doi: 10.1016/j.jvs.2012.07.051. Epub 2012 Oct 6. PMID 23044259
- [Background] Pande RL, Perlstein TS, Beckman JA, Creager MA. Secondary prevention and mortality in peripheral artery disease: National Health and Nutrition Examination Study, 1999 to 2004. Circulation. 2011 Jul 5;124(1):17-23. doi: 10.1161/CIRCULATIONAHA.110.003954. Epub 2011 Jun 20. PMID 21690489
- [Background] Nordanstig J, Broeren M, Hensater M, Perlander A, Osterberg K, Jivegard L. Six-minute walk test closely correlates to "real-life" outdoor walking capacity and quality of life in patients with intermittent claudication. J Vasc Surg. 2014 Aug;60(2):404-9. doi: 10.1016/j.jvs.2014.03.003. Epub 2014 Mar 29. PMID 24690492
- [Background] Colas-Ribas C, Signolet I, Henni S, Feuillloy M, Gagnadoux F, Abraham P. High prevalence of known and unknown pulmonary diseases in patients with claudication during exercise oximetry: A retrospective analysis. Medicine (Baltimore). 2016 Oct;95(40):e4888. doi: 10.1097/MD.0000000000004888. PMID 27749546
- [Background] Sieminski DJ, Gardner AW. The relationship between free-living daily physical activity and the severity of peripheral arterial occlusive disease. Vasc Med. 1997 Nov;2(4):286-91. doi: 10.1177/1358863X9700200402. PMID 9575600
- [Background] Gardner AW, Montgomery PS, Scott KJ, Blevins SM, Afaq A, Nael R. Association between daily ambulatory activity patterns and exercise performance in patients with intermittent claudication. J Vasc Surg. 2008 Nov;48(5):1238-44. doi: 10.1016/j.jvs.2008.06.062. Epub 2008 Sep 4. PMID 18771878